CLINICAL TRIAL: NCT04456673
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, 52-week Pivotal Study to Assess the Efficacy, Safety, and Tolerability of Dupilumab in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD) With Type 2 Inflammation
Brief Title: Pivotal Study to Assess the Efficacy, Safety and Tolerability of Dupilumab in Patients With Moderate to Severe COPD With Type 2 Inflammation
Acronym: NOTUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15805; U1111-1211-8837 (Registry Identifier: ICTRP); 2018-001954-91 (EudraCT Number)
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Participants received dupilumab 300 mg subcutaneous (SC) injection every 2 weeks (q2w) up to 52 weeks
  Interventions: Drug: Dupilumab SAR231893; Drug: Inhaled Corticosteroid; Drug: Inhaled Long-Acting Beta Agonist; Drug: Inhaled Long-Acting Muscarinic Antagonist
- Placebo (Placebo Comparator): Participants received placebo matched to dupilumab 300 mg SC injection q2w up to 52 weeks
  Interventions: Drug: Inhaled Corticosteroid; Drug: Inhaled Long-Acting Beta Agonist; Drug: Inhaled Long-Acting Muscarinic Antagonist; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Inhaled Corticosteroid — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Inhaled Long-Acting Beta Agonist — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Inhaled Long-Acting Muscarinic Antagonist — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab administered every 2 weeks in patients with moderate or severe Chronic Obstructive Pulmonary Disease (COPD) as measured by

* Annualized rate of acute moderate or severe COPD exacerbation (AECOPD)

Secondary Objectives:

To evaluate the effect of dupilumab administered every 2 weeks on

* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) over 12 weeks compared to placebo
* Health related quality of life, assessed by the change from baseline to Week 52 in the St. George's Respiratory Questionnaire (SGRQ)
* Pre-bronchodilator FEV1 over 52 weeks compared to placebo
* Lung function assessments
* Moderate and severe COPD exacerbations
* To evaluate safety and tolerability
* To evaluate dupilumab systemic exposure and incidence of antidrug antibodies (ADA)

DETAILED DESCRIPTION:
Approximately 68 weeks including a 4-week screening period, a 52-week treatment period, and 12 weeks of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Participants with a physician diagnosis of COPD who met the following criteria at screening:

  * Current or former smokers with a smoking history of ≥10 pack-years.
  * Moderate-to-severe COPD (post-bronchodilator FEV1/ forced vital capacity [FVC] ratio <0.70 and post-bronchodilator FEV1 % predicted >30% and ≤70%).
  * Medical Research Council (MRC) Dyspnea Scale grade ≥2.
  * Patient-reported history of signs and symptoms of chronic bronchitis (chronic productive cough) for 3 months in the year up to screening in the absence of other known causes of chronic cough.
  * Documented history of high exacerbation risk defined as exacerbation history of ≥2 moderate or ≥1 severe within the year prior to inclusion. At least one exacerbation should have occurred while the participant was taking inhaled corticosteroid (ICS)/long-acting beta agonist (LABA)/long-acting muscarinic antagonist (LAMA) (or LABA/LAMA if ICS is contraindicated). Moderate exacerbations were recorded by the investigator and defined as AECOPD that required either systemic corticosteroids (intramuscular, intravenous, or oral) and/or antibiotics. One of the two required moderate exacerbations had to require the use of systemic corticosteroids. Severe exacerbations were recorded by the investigator and defined as AECOPD requiring hospitalization or observation > 24 hours in emergency department/urgent care facility.
  * Background triple therapy (ICS + LABA + LAMA) for 3 months prior to randomization with a stable dose of medication for ≥1 month prior to Visit 1; Double therapy (LABA + LAMA) allowed if ICS is contraindicated.
* Evidence of Type 2 inflammation: Participants with blood eosinophils ≥300 cells/microliter at Visit 1.

Exclusion Criteria:

* COPD diagnosis for less than 12 months prior to randomization.
* Participants with current diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines, or documented history of asthma.
* Significant pulmonary disease other than COPD (e.g., lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome etc) or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* Cor pulmonale, evidence of right cardiac failure.
* Long-term treatment with oxygen >4.0 L/min OR if a participant requires more than 2.0 L/min in order to maintain oxygen saturation >88%
* Hypercapnia requiring Bi-level ventilation.
* AECOPD as defined in inclusion criteria within 4 weeks prior to screening, or during the screening period.
* Respiratory tract infection within 4 weeks prior to screening, or during the screening period.
* History of, or planned pneumonectomy or lung volume reduction surgery. Participants who were participating in the acute phase of a pulmonary rehabilitation program, ie, who started rehabilitation <4 weeks prior to screening (Note: participants in the maintenance phase of a rehabilitation program can be included).
* Diagnosis of α-1 anti-trypsin deficiency.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 935 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (334):
- United States (92):
  - Cullman Research Center, LLC Site Number : 8400095, Cullman, Alabama
  - Pulmonary & Sleep Associates of Jasper PC Site Number : 8400090, Jasper, Alabama
  - Scottsboro Quick Care Clinic Site Number : 8400116, Scottsboro, Alabama
  - Phoenix Medical Group Site Number : 8400061, Peoria, Arizona
  - Medical Advancement Center of Arizona Site Number : 8400107, Tempe, Arizona
  - Asthma and Allergy Institute Site Number : 8400022, Little Rock, Arkansas
  - Kern Research, Inc Site Number : 8400031, Bakersfield, California
  - NewportNativeMD, Inc Site Number : 8400032, Newport Beach, California
  - Prospective Research Innovations, Inc. Site Number : 8400063, Rancho Cucamonga, California
  - ACRC Studies Site Number : 8400094, San Diego, California
  - Institute of HealthCare Assessment, Inc. Site Number : 8400015, San Diego, California
  - Allianz Research Institute Site Number : 8400007, Westminster, California
  - Innovative Clinical Research Site Number : 8400018, Lafayette, Colorado
  - Helix Biomedics, LLC Site Number : 8400035, Boynton Beach, Florida
  - Pioneer Clinical Research Site Number : 8400043, Boynton Beach, Florida
  - Renaissance Research and Medical Group, Inc Site Number : 8400092, Cape Coral, Florida
  - St. Francis Sleep, Allergy and Lung Institute Site Number : 8400020, Clearwater, Florida
  - Beautiful Minds Clinical Research Center Site Number : 8400081, Cutler Bay, Florida
  - Omega Research Consultants, LLC Site Number : 8400021, DeBary, Florida
  - Sciences Connections, LLC Site Number : 8400133, Doral, Florida
  - InvesClinic, LLC Site Number : 8400039, Fort Lauderdale, Florida
  - Finlay Medical Research Site Number : 8400071, Greenacres City, Florida
  - Direct Helpers Medical Center Inc Site Number : 8400079, Hialeah, Florida
  - DL Research Solutions Inc Site Number : 8400089, Miami, Florida
  - Phoenix Medical Research, LLC Site Number : 8400012, Miami, Florida
  - Columbus Clinical Services Site Number : 8400062, Miami, Florida
  - Reed Medical Research Site Number : 8400123, Miami, Florida
  - De La Cruz Research Center, LLC Site Number : 8400075, Miami, Florida
  - Florida Institute for Clinical Research Site Number : 8400129, Orlando, Florida
  - Central Florida Pulmonary Group, PA Site Number : 8400101, Orlando, Florida
  - Innovation Medical Research Center Site Number : 8400114, Palmetto Bay, Florida
  - Family Medical Specialists of Florida, PA Site Number : 8400077, Plant City, Florida
  - Coastal Pulmonary And Critical Care Site Number : 8400013, St. Petersburg, Florida
  - Florida Pulmonary Research Center Site Number : 8400001, Winter Park, Florida
  - Appalachian Clinical Research Site Number : 8400048, Adairsville, Georgia
  - Northlake Medical Group Site Number : 8400099, Atlanta, Georgia
  - River Birch Research, LLC Site Number : 8400045, Blue Ridge, Georgia
  - Medical Centre of Conyers Site Number : 8400064, Conyers, Georgia
  - David Kavtaradze MD, Inc. Site Number : 8400135, Cordele, Georgia
  - Gwinnett Biomedical Research Site Number : 8400052, Lawrenceville, Georgia
  - Southeast Lung Associates Site Number : 8400003, Rincon, Georgia
  - Herman Clinical Research LLC Site Number : 8400078, Suwanee, Georgia
  - Avant Research Associates LLC Site Number : 8400118, Crowley, Louisiana
  - Genesis Clinical Research & Consulting Site Number : 8400050, Fall River, Massachusetts
  - Infinity Medical Research Site Number : 8400004, South Dartmouth, Massachusetts
  - Henry Ford Health System Site Number : 8400053, Detroit, Michigan
  - Revive Research Institute Site Number : 8400120, Lathrup Village, Michigan
  - Romedica, LLC Site Number : 8400034, Rochester, Michigan
  - Covenant Healthcare Site Number : 8400057, Saginaw, Michigan
  - Great Lakes Research Institute Site Number : 8400096, Southfield, Michigan
  - Montana Medical Research Site Number : 8400019, Missoula, Montana
  - Somnos Clinical Research Site Number : 8400016, Lincoln, Nebraska
  - Quality Clinical Research, Inc. Site Number : 8400073, Omaha, Nebraska
  - Jersey City Breathing Center Site Number : 8400137, Jersey City, New Jersey
  - WellNow Urgent Care Site Number : 8400132, East Amherst, New York
  - Northwell Health Site Number : 8400054, New Hyde Park, New York
  - Mid Hudson Medical Research PLLC Site Number : 8400037, New Windsor, New York
  - Great Lakes Medical Research Site Number : 8400044, Westfield, New York
  - Onsite Clinical Solutions LLC Site Number : 8400042, Charlotte, North Carolina
  - Clinical Research of Gastonia Site Number : 8400010, Gastonia, North Carolina
  - Monroe Biomedical Research Site Number : 8400087, Monroe, North Carolina
  - Lake Norman Pulmonary and Sleep Medicine - Mooresville Site Number : 8400006, Mooresville, North Carolina
  - Lapis Clinical Research At BlueSkies Family Medicine Site Number : 8400117, Mooresville, North Carolina
  - Coastal Carolina Health Care, P.A. Site Number : 8400025, New Bern, North Carolina
  - Southeastern Research Center Site Number : 8400068, Winston-Salem, North Carolina
  - Optimed Research, LTD Site Number : 8400082, Columbus, Ohio
  - Toledo Institute of Clinical Research Site Number : 8400024, Toledo, Ohio
  - Allergy, Asthma and Clinical Research Center Site Number : 8400127, Oklahoma City, Oklahoma
  - Clinical Research of Central PA Site Number : 8400009, DuBois, Pennsylvania
  - Frontier Clinical Research, LLC Site Number : 8400049, Scottdale, Pennsylvania
  - Carolina Medical Research, LLC Site Number : 8400026, Clinton, South Carolina
  - MD First Research Site Number : 8400105, Lancaster, South Carolina
  - LLM Research Site Number : 8400125, Myrtle Beach, South Carolina
  - Health Concepts Site Number : 8400027, Rapid City, South Dakota
  - Pulmonary & Sleep Specialists Site Number : 8400136, Dickson, Tennessee
  - Clinical Trials Center of Middle Tennessee Site Number : 8400066, Franklin, Tennessee
  - MultiSpecialty Clinical Research Site Number : 8400110, Johnson City, Tennessee
  - REX Clinical Trials Site Number : 8400143, Beaumont, Texas
  - Clinrx Research Site Number : 8400059, Carrollton, Texas
  - Houston Pulmonary and Sleep Associates Site Number : 8400011, Cypress, Texas
  - Biopharma Informatic - Cardiff Avenue - PPDS Site Number : 8400055, Houston, Texas
  - Prolato Clinical Research Center Site Number : 8400128, Houston, Texas
  - Pioneer Research Solutions, Inc. Site Number : 8400070, Houston, Texas
  - Radiance Clinical Research Site Number : 8400029, Lampasas, Texas
  - DCOL Center for Clinical Research Site Number : 8400028, Longview, Texas
  - Metroplex Pulmonary and Sleep Center Site Number : 8400131, McKinney, Texas
  - Clinrx Research, LLC Site Number : 8400069, Plano, Texas
  - Diagnostics Research Group Site Number : 8400038, San Antonio, Texas
  - Mt. Olympus Medical Research Site Number : 8400115, Sugar Land, Texas
  - Pulmonary Research of Abingdon, LLC Site Number : 8400030, Abingdon, Virginia
  - Clinical Research Partners Site Number : 8400040, Richmond, Virginia
  - Allergy, Asthma & Sinus Center, S.C. Site Number : 8400088, Greenfield, Wisconsin
- Argentina (13):
  - Investigational Site Number : 0320007, Berazategui, Buenos Aires
  - Investigational Site Number : 0320006, CABA, Buenos Aires
  - Investigational Site Number : 0320004, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320010, La Plata, Buenos Aires
  - Investigational Site Number : 0320013, Lobos, Buenos Aires
  - Investigational Site Number : 0320005, Quilmes, Buenos Aires F.D.
  - Investigational Site Number : 0320011, Córdoba, Córdoba Province
  - Investigational Site Number : 0320008, Rosario, Santa Fe Province
  - Investigational Site Number : 0320009, Rosario, Santa Fe Province
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320012, Launs Este
- Australia (3):
  - Investigational Site Number : 0360008, Kent Town, South Australia
  - Investigational Site Number : 0360005, Clayton, Victoria
  - Investigational Site Number : 0360001, Spearwood, Western Australia
- Belgium (4):
  - Investigational Site Number : 0560002, Edegem
  - Investigational Site Number : 0560001, Leuven
  - Investigational Site Number : 0560003, Liège
  - Investigational Site Number : 0560004, Mechelen
- Brazil (14):
  - CEDOES - Centro de Diagnostico e Pesquisa de Osteoporose do ES Site Number : 0760020, Vitória, Espírito Santo
  - SER da Bahia Site Number : 0760019, Salvador, Estado de Bahia
  - Instituto Mederi de Pesquisa e Saude Site Number : 0760008, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre Site Number : 0760017, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - HOSPITAL DIA DO PULMAO Site Number : 0760006, Blumenau, Santa Catarina
  - UFSC - Hospital Universitário Site Number : 0760018, Florianópolis, Santa Catarina
  - PUC Campinas - Sociedade Campineira de Educaçao e Instruçao Site Number : 0760015, Campinas, São Paulo
  - FUNDACAO DO ABC - FACULDADE DE MEDICINA DO ABC (FMABC) Site Number : 0760007, Santo André, São Paulo
  - CPQuali Pesquisa Clinica Site Number : 0760003, São Paulo, São Paulo
  - Instituto de Pesquisa Grupo NotreDame Intermedica Site Number : 0760012, São Paulo, São Paulo
  - Nucleo de Pesquisa Clinica e Ensino da Rede Sao Camilo Site Number : 0760021, São Paulo, São Paulo
  - InCor - Instituto do Coraçao do Hospital das Clinicas da FMUSP Site Number : 0760002, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila Site Number : 0760009, Sorocaba, São Paulo
- Bulgaria (19):
  - Investigational Site Number : 1005025, Burgas
  - Investigational Site Number : 1005021, Dupnitsa
  - Investigational Site Number : 1005012, Haskovo
  - Investigational Site Number : 1005011, Montana
  - Investigational Site Number : 1005008, Plovdiv
  - Investigational Site Number : 1005015, Rousse
  - Investigational Site Number : 1005013, Rousse
  - Investigational Site Number : 1005018, Sofia
  - Investigational Site Number : 1005003, Sofia
  - Investigational Site Number : 1005001, Sofia
  - Investigational Site Number : 1005006, Sofia
  - Investigational Site Number : 1005002, Sofia
  - Investigational Site Number : 1005026, Sofia
  - Investigational Site Number : 1005024, Stara Zagora
  - Investigational Site Number : 1005004, Stara Zagora
  - Investigational Site Number : 1005023, Veliko Tyrnovo
  - Investigational Site Number : 1005027, Veliko Tyrnovo
  - Investigational Site Number : 1005019, Vidin
  - Investigational Site Number : 1005020, Vratsa
- Canada (11):
  - Investigational Site Number : 1240015, Calgary, Alberta
  - Investigational Site Number : 1240018, Kamloops, British Columbia
  - Investigational Site Number : 1240017, Kelowna, British Columbia
  - Investigational Site Number : 1240014, Moncton, New Brunswick
  - Investigational Site Number : 1240010, Ajax, Ontario
  - Investigational Site Number : 1240009, Sarnia, Ontario
  - Investigational Site Number : 1240007, Windsor, Ontario
  - Investigational Site Number : 1240004, Montreal, Quebec
  - Investigational Site Number : 1240012, Québec, Quebec
  - Investigational Site Number : 1240001, Québec
  - Investigational Site Number : 1240005, Québec
- Chile (7):
  - Investigational Site Number : 1520009, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520006, Curicó, Maule Region
  - Investigational Site Number : 1520001, Talca, Maule Region
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Quillota, Región de Valparaíso
- Colombia (3):
  - Investigational Site Number : 1700002, Bogotá
  - Investigational Site Number : 1700007, Bucaramanga
  - Investigational Site Number : 1700005, Manizales
- Czechia (7):
  - Investigational Site Number : 2030009, Havlíčkův Brod
  - Investigational Site Number : 2030004, Jihlava
  - Investigational Site Number : 2030001, Jindrichuv Hradec III
  - Investigational Site Number : 2030007, Kralupy nad Vltavou
  - Investigational Site Number : 2030003, Miroslav
  - Investigational Site Number : 2030010, Nymburk
  - Investigational Site Number : 2030002, Strakonice
- France (8):
  - Investigational Site Number : 2500009, Bayonne
  - Investigational Site Number : 2500002, Dijon
  - Investigational Site Number : 2500005, Lyon
  - Investigational Site Number : 2500003, Montpellier
  - Investigational Site Number : 2500007, Paris
  - Investigational Site Number : 2500008, Paris
  - Investigational Site Number : 2500006, Pessac
  - Investigational Site Number : 2500001, Saint-Herblain
- Germany (15):
  - Investigational Site Number : 2760024, Berlin
  - Investigational Site Number : 2760025, Berlin
  - Investigational Site Number : 2760017, Darmstadt
  - Investigational Site Number : 2760009, Frankfurt am Main
  - Investigational Site Number : 2760002, Hamburg
  - Investigational Site Number : 2760003, Hanover
  - Investigational Site Number : 2760007, Koblenz
  - Investigational Site Number : 2760023, Leipzig
  - Investigational Site Number : 2760011, Leipzig
  - Investigational Site Number : 2760010, Lübeck
  - Investigational Site Number : 2760012, Mainz
  - Investigational Site Number : 2760008, Marburg
  - Investigational Site Number : 2760020, Peine
  - Investigational Site Number : 2760016, Rosenheim
  - Investigational Site Number : 2760018, Wiesbaden
- Greece (6):
  - Investigational Site Number : 3000006, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Heraklion
  - Investigational Site Number : 3000002, Ioannina
  - Investigational Site Number : 3000007, Palaio Faliro, Athens
  - Investigational Site Number : 3000004, Thessaloniki
- Hungary (6):
  - Investigational Site Number : 3480003, Edelény
  - Investigational Site Number : 3480004, Gödöllö
  - Investigational Site Number : 3480002, Hajdunánás
  - Investigational Site Number : 3480006, Mosonmagyaróvár
  - Investigational Site Number : 3480001, Százhalombatta
  - Investigational Site Number : 3480005, Szombathely
- Latvia (7):
  - Investigational Site Number : 4280008, Balvi
  - Investigational Site Number : 4280007, Rēzekne
  - Investigational Site Number : 4280001, Riga
  - Investigational Site Number : 4280005, Riga
  - Investigational Site Number : 4280006, Riga
  - Investigational Site Number : 4280002, Riga
  - Investigational Site Number : 4280003, Riga
- Lithuania (5):
  - Investigational Site Number : 4400001, Kaunas
  - Investigational Site Number : 4400003, Kaunas
  - Investigational Site Number : 4400008, Kaunas
  - Investigational Site Number : 4400007, Klaipėda
  - Investigational Site Number : 4400005, Vilnius
- Mexico (11):
  - Investigational Site Number : 4840002, Guadalajara, Jalisco
  - Investigational Site Number : 4840013, Guadalajara, Jalisco
  - Investigational Site Number : 4840011, Zapopan, Jalisco
  - Investigational Site Number : 4840008, Benito Juárez, Mexico City
  - Investigational Site Number : 4840004, Monterrey, Nuevo León
  - Investigational Site Number : 4840003, Monterrey, Nuevo León
  - Investigational Site Number : 4840010, Chihuahua City
  - Investigational Site Number : 4840006, Durango
  - Investigational Site Number : 4840007, Mexico City
  - Investigational Site Number : 4840009, Mexico City
  - Investigational Site Number : 4840005, Veracruz
- Netherlands (9):
  - Investigational Site Number : 5280005, Arnhem
  - Investigational Site Number : 5280001, Breda
  - Investigational Site Number : 5280010, Dordrecht
  - Investigational Site Number : 5280009, Harderwijk
  - Investigational Site Number : 5280002, Leeuwarden
  - Investigational Site Number : 5280006, Nijmegen
  - Investigational Site Number : 5280011, Roermond
  - Investigational Site Number : 5280008, Zutphen
  - Investigational Site Number : 5280004, Zwolle
- Peru (5):
  - Investigational Site Number : 6040006, Lima
  - Investigational Site Number : 6040004, Lima
  - Investigational Site Number : 6040001, Lima
  - Investigational Site Number : 6040002, Lima Lima
  - Investigational Site Number : 6040005, Piura
- Poland (11):
  - Investigational Site Number : 6160009, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160007, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160015, Grodzisk Mazowiecki, Masovian Voivodeship
  - Investigational Site Number : 6160010, Rzeszów, Podkarpackie Voivodeship
  - Investigational Site Number : 6160008, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160018, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160011, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160014, Elblag, Warmian-Masurian Voivodeship
  - Investigational Site Number : 6160019, Krakow
  - Investigational Site Number : 6160020, Nowa Sól
  - Investigational Site Number : 6160022, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Portugal (5):
  - Investigational Site Number : 6200007, Almada
  - Investigational Site Number : 6200006, Aveiro
  - Investigational Site Number : 6200002, Guimarães
  - Investigational Site Number : 6200009, Lisbon
  - Investigational Site Number : 6200012, Matosinhos Municipality
- Romania (6):
  - Investigational Site Number : 6425004, Bacau
  - Investigational Site Number : 6425003, Cluj-Napoca
  - Investigational Site Number : 6425005, Constanța
  - Investigational Site Number : 6425002, Iași
  - Investigational Site Number : 6425006, Piteşti
  - Investigational Site Number : 6425001, Timișoara
- Russia (12):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430003, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430009, Nizhny Novgorod
  - Investigational Site Number : 6430010, Ryazan
  - Investigational Site Number : 6430004, Saint Petersburg
  - Investigational Site Number : 6430013, Saint Petersburg
  - Investigational Site Number : 6430014, Saint Petersburg
  - Investigational Site Number : 6430012, Stavropol
  - Investigational Site Number : 6430006, Tomsk
  - Investigational Site Number : 6430008, Ulyanovsk
  - Investigational Site Number : 6430005, Voronezh
- Serbia (6):
  - Investigational Site Number : 6880005, Belgrade
  - Investigational Site Number : 6880006, Belgrade
  - Investigational Site Number : 6880007, Belgrade
  - Investigational Site Number : 6880001, Kamenitz
  - Investigational Site Number : 6880003, Kragujevac
  - Investigational Site Number : 6880002, Valjevo
- Slovakia (6):
  - Investigational Site Number : 7030007, Banská Bystrica
  - Investigational Site Number : 7030006, Humenné
  - Investigational Site Number : 7030005, Košice
  - Investigational Site Number : 7030003, Levice
  - Investigational Site Number : 7030001, Poprad
  - Investigational Site Number : 7030002, Spišská Nová Ves
- South Africa (14):
  - Investigational Site Number : 7100015, Benoni
  - Investigational Site Number : 7100004, Cape Town
  - Investigational Site Number : 7100014, Chatsworth
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100013, Durban
  - Investigational Site Number : 7100003, Durban
  - Investigational Site Number : 7100010, Durban
  - Investigational Site Number : 7100002, Gatesville
  - Investigational Site Number : 7100011, Gauteng
  - Investigational Site Number : 7100009, Johannesburg
  - Investigational Site Number : 7100012, Middelburg
  - Investigational Site Number : 7100006, Parow
  - Investigational Site Number : 7100005, Pretoria
  - Investigational Site Number : 7100008, Somerset West
- Spain (8):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240009, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240012, Cáceres, Cáceres
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240007, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240008, Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7240010, Málaga
  - Investigational Site Number : 7240011, Zaragoza
- Ukraine (10):
  - Investigational Site Number : 8040011, Chernivtsi
  - Investigational Site Number : 8040002, Ivano-Frankivsk
  - Investigational Site Number : 8040003, Ivano-Frankivsk
  - Investigational Site Number : 8040001, Kharkiv
  - Investigational Site Number : 8040007, Kyiv
  - Investigational Site Number : 8040004, Kyiv
  - Investigational Site Number : 8040006, Lviv
  - Investigational Site Number : 8040010, Ternopil
  - Investigational Site Number : 8040008, Zaporizhzhia
  - Investigational Site Number : 8040009, Zaporizhzhya
- United Kingdom (11):
  - Investigational Site Number : 8260003, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260002, Blackpool, Lancashire
  - Investigational Site Number : 8260006, Swansea, Neath Port Talbot
  - Investigational Site Number : 8260007, North Shields, Newcastle Upon Tyne
  - Investigational Site Number : 8260004, South Shields, Newcastle Upon Tyne
  - Investigational Site Number : 8260013, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260012, Aylesbury
  - Investigational Site Number : 8260001, Bradford
  - Investigational Site Number : 8260005, Bristol
  - Investigational Site Number : 8260011, Chippenham
  - Investigational Site Number : 8260015, Derby

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Bhatt SP, Rabe KF, Hanania NA, Vogelmeier CF, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Dakin P, Maloney J, Lu X, Bauer D, Bansal A, Abdulai RM, Robinson LB. Effect of Dupilumab on Health-Related Quality of Life and Respiratory Symptoms in Patients With COPD and Type 2 Inflammation: BOREAS and NOTUS. Chest. 2025 Jul;168(1):56-66. doi: 10.1016/j.chest.2025.01.029. Epub 2025 Jan 31. PMID 39894389
- [Derived] Bhatt SP, Rabe KF, Hanania NA, Vogelmeier CF, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Patel N, Yancopoulos GD, Akinlade B, Maloney J, Lu X, Bauer D, Bansal A, Abdulai RM, Robinson LB; NOTUS Study Investigators. Dupilumab for COPD with Blood Eosinophil Evidence of Type 2 Inflammation. N Engl J Med. 2024 Jun 27;390(24):2274-2283. doi: 10.1056/NEJMoa2401304. Epub 2024 May 20. PMID 38767614
- See also: EFC15805 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25232&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 329 centers in 29 countries. A total of 2769 participants were screened between 06 July 2020 to 19 April 2023, of which 1834 participants were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 935 participants were randomized in a 1:1 ratio to receive either dupilumab 300 milligrams (mg) every 2 weeks (q2w) or matching placebo. Randomization was stratified by country, inhaled corticosteroid (ICS) dose (high-dose ICS [yes/no]) at baseline, and smoking status at screening (current smokers or not).
Groups:
- Placebo: Participants received placebo matched to dupilumab 300 mg subcutaneous (SC) injection q2w up to 52 weeks.
- Dupilumab 300 mg q2w: Participants received dupilumab 300 mg SC injection q2w up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w
Started (Randomized) | 465 | 470
Randomized and Treated | 465 | 468
Safety Population (1 participant was exposed to different treatment other than planned (was allocated to placebo arm but inadvertently received dupilumab 300 mg q2w on Day 113). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.) | 464 | 469
Completed | 422 | 428
Not Completed | 43 | 42
Not completed — Adverse Event | 7 | 14
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Withdrawal by Subject | 31 | 23
Not completed — Not related to Coronavirus Disease-2019 (COVID-19) | 4 | 5

BASELINE CHARACTERISTICS:
Population: The Randomized population included all participants who had been allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 465 | 470 | 935
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (8.5) | 65.2 (8.1) | 65.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 150 | 303
  Male | 312 | 320 | 632
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 26 | 22 | 48
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 4 | 12
  White | 416 | 422 | 838
  More than one race | 8 | 12 | 20
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Over the 52-week Treatment Period
Description: Moderate exacerbations were recorded by the Investigator and defined as acute exacerbation of COPD (AECOPD) event that required either systemic corticosteroids (such as intramuscular, intravenous, or oral) and/or antibiotics. Severe exacerbations were also recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Annualized event rate was the total number of events that occurred during the 52-week treatment period divided by the total number of participant-years followed in the 52-week treatment period.
Time Frame: Baseline (Day 1) to Week 52
Population: The Intent-to-treat (ITT) population included all randomized participants analyzed according to the treatment group allocated by randomization.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 465 | 470
Exacerbation per participant-year | 1.295 [1.048 to 1.600] | 0.859 [0.699 to 1.057]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived using negative binomial model with the total number of the events occurring during the 52-week treatment period as the response variable, and treatment group, region (pooled country), ICS dose, smoking status at screening, baseline disease severity, and number of moderate or severe COPD exacerbation events within one year prior to the study as covariates, and log-transformed treatment duration as an offset variable; Test type: Superiority — A hierarchical testing procedure was used to control type I error and handle primary and first 4 secondary endpoints (reported sequentially) analyses at a 2-sided significance level of 0.05; p = 0.0002, Negative binomial model; Risk Difference (RD) = -0.435, 95% CI 2-sided [-0.682 to -0.188] — Derived using delta method

2. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) to Week 12
Description: The FEV1 was defined as the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Spirometry was performed after a wash out period of bronchodilators according to their action duration. Baseline was defined as the last available value up to randomization but prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Week 12
Population: The ITT population included all randomized participants analyzed according to the treatment group allocated by randomization. Only those participants with data collected are reported.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 461 | 464
Liters | 0.057 (0.017) | 0.139 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from mixed-effect model with repeated measures (MMRM) model with the change from baseline in pre-bronchodilator FEV1 up to Week 12 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-bronchodilator FEV1, and FEV1 baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0001, MMRM model; Least Square (LS) Mean Difference = 0.082, 95% CI 2-sided [0.040 to 0.124]

3. Secondary Outcome: Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Total Score to Week 52
Description: The SGRQ is a 50-item self-administered questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation and rated on electronic diary. Scores by dimension were calculated for 3 domains: symptoms (respiratory symptoms: frequency and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response had a unique empirically derived weight where lowest possible weight was 0 and the highest was 100. Total score was obtained by summing all positive responses in the questionnaire. The total score and domain score was derived from the relevant items and converted to a score of 0 to 100 with a higher score indicating worse health status/health related quality of life. Baseline was defined as the last available value up to randomization but prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population with an opportunity to reach Week 52 included participants who had an opportunity to reach Week 52 assessments and were analyzed for the continuous and proportion type endpoints at Week 52. Only those participants with data collected are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 342 | 350
score on a scale | -6.444 (0.922) | -9.816 (0.920)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in SGRQ total score up to Week 52 as response variables, and treatment group, region (pooled country), ICS dose, smoking status at screening, treatment-by-visit interaction, baseline SGRQ total score, and SGRQ baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0068, MMRM model; LS Mean Difference = -3.371, 95% CI 2-sided [-5.811 to -0.931]

4. Secondary Outcome: Percentage of Participants With Saint George's Respiratory Questionnaire Improvement ≥4 Points at Week 52
Description: A responder was defined as a participant with improvement from baseline in SGRQ total score at Week 52 by ≥4 points. Percentage of participants who achieved a clinically meaningful response in SGRQ total score (improvement by ≥4 points)/responders are reported. SGRQ is a 50-item self-administered questionnaire. Scores by dimension were calculated for 3 domains: symptoms (respiratory symptoms: frequency and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response had unique empirically derived weight where lowest possible weight was 0 and highest was 100. Total score was obtained by summing all positive responses in questionnaire. Total score and domain score was derived from relevant items and converted to a score of 0 to 100; higher score indicating worse health status/health related quality of life.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population with an opportunity to reach Week 52 included participants who had an opportunity to reach Week 52 assessments and were analyzed for the continuous and proportion type endpoints at Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 359 | 362
Percentage of participants | 46.5 | 51.4
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from logistic regression model which includes treatment group, region (pooled country), ICS dose, smoking status at screening, and baseline SGRQ total score as covariates; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3329, Regression, Logistic; Odds Ratio (OR) = 1.164, 95% CI 2-sided [0.856 to 1.581]

5. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second to Week 52
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 356 | 359
Liters | 0.054 (0.020) | 0.115 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in pre-bronchodilator FEV1 up to Week 52 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-bronchodilator FEV1, and FEV1 baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0182, MMRM model; LS Mean Difference = 0.062, 95% CI 2-sided [0.011 to 0.113]

6. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second to Weeks 2, 4, 8, 24, 36, and 44
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 24, 36 and 44
Population: The ITT population with an opportunity to reach Week 52 included participants who had an opportunity to reach Week 52 assessments and were analyzed for all weeks up to Week 52. Only those participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 356 | 359
Liters
  Week 2 | 0.072 (0.018) | 0.108 (0.018)
  Week 4 | 0.077 (0.018) | 0.132 (0.019)
  Week 8 | 0.069 (0.019) | 0.133 (0.020)
  Week 24 | 0.064 (0.020) | 0.154 (0.021)
  Week 36 | 0.068 (0.021) | 0.117 (0.021)
  Week 44 | 0.065 (0.020) | 0.154 (0.021)

7. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in 1 Second to Weeks 2, 4, 8, 12, 24, 36, and 52
Description: The FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Post-bronchodilator FEV1 referred to the spirometry performed consistent with the mechanism of action of reliever (30 minutes for albuterol or another short-acting beta agonists). Baseline was defined as the last available value up to randomization but prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 356 | 358
Liters
  Week 2 | 0.082 (0.018) | 0.101 (0.018)
  Week 4 | 0.098 (0.018) | 0.126 (0.018)
  Week 8 | 0.083 (0.019) | 0.147 (0.020)
  Week 12 | 0.064 (0.020) | 0.136 (0.020)
  Week 24 | 0.081 (0.020) | 0.152 (0.020)
  Week 36 | 0.070 (0.020) | 0.131 (0.021)
  Week 52 | 0.059 (0.020) | 0.127 (0.021)

8. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) 25 to 75 Percent (%) to Weeks 2, 4, 8, 12, 24, 36, 44, and 52
Description: FEF is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF 25-75% was defined as the FEF at 25% to 75% of forced vital capacity (FVC), where FVC was defined as the volume of air that can be forcibly blown out after full inspiration in the upright position. Spirometry was performed after a wash out period of bronchodilators according to their action duration. Baseline was defined as the last available value up to randomization but prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 24, 36, 44 and 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters per second
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 356 | 359
Liters per second
  Week 2 | 0.057 (0.018) | 0.103 (0.018)
  Week 4 | 0.056 (0.018) | 0.114 (0.018)
  Week 8 | 0.059 (0.019) | 0.134 (0.019)
  Week 12 | 0.066 (0.021) | 0.137 (0.021)
  Week 24 | 0.051 (0.019) | 0.147 (0.020)
  Week 36 | 0.073 (0.021) | 0.128 (0.022)
  Week 44 | 0.053 (0.021) | 0.154 (0.021)
  Week 52 | 0.065 (0.020) | 0.122 (0.020)

9. Secondary Outcome: Annualized Rate of Severe Chronic Obstructive Pulmonary Disease Exacerbations Over the 52-week Treatment Period
Description: Severe exacerbations were recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Annualized event rate was the total number of events that occurred during the 52-week treatment period divided by the total number of participant-years followed in the 52-week treatment period.
Time Frame: Baseline (Day 1) to Week 52
Population: The ITT population included all randomized participants analyzed according to the treatment group allocated by randomization.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 465 | 470
Exacerbation per participant-year | 0.124 [0.072 to 0.215] | 0.070 [0.039 to 0.123]

10. Secondary Outcome: Time to First Moderate or Severe Chronic Obstructive Pulmonary Disease Exacerbation Event During the 52-week Treatment Period
Description: The time to first moderate or severe exacerbation was defined as date of the first event minus randomization date +1. Moderate exacerbations were recorded by the Investigator and defined as AECOPD event that required either systemic corticosteroids (such as intramuscular, intravenous, or oral) and/or antibiotics. Severe exacerbations were recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Median time as well as 95% confidence interval was calculated using Kaplan-Meier estimates.
Time Frame: Baseline (Day 1) and up to Weeks 12, 24, 36 and 52
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 465 | 470
Weeks
  Week 12 | 0.172 [0.139 to 0.207] | 0.108 [0.081 to 0.138]
  Week 24 | 0.265 [0.225 to 0.306] | 0.206 [0.170 to 0.244]
  Week 36 | 0.342 [0.298 to 0.387] | 0.292 [0.250 to 0.335]
  Week 52 | 0.424 [0.375 to 0.471] | 0.361 [0.315 to 0.407]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed or worsened or became serious during TE period (between the first administration of study treatment to the last administration of the study treatment + 98 days).
Time Frame: From the first dose of study treatment (Day 1) up to the last dose of the study treatment + 98 days, up to 506 days
Population: The Safety population included all participants who actually received at least 1 dose or partial of a dose of the study treatment, analyzed according to the treatment participants actually received. 1 participant was exposed to different treatment other than planned (was allocated to placebo arm but inadvertently received dupilumab 300 mg q2w on Day 113). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 464 | 469
Participants
  Any TEAE | 330 | 322
  Any TESAE | 79 | 65

12. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Hematology
Description: Blood samples were collected to determine PCSA in hematology. PCSA values were defined as abnormal values considered medically important by the Sponsor according to pre-defined criteria/thresholds based on literature review and defined by the Sponsor for clinical laboratory tests. Criteria for PCSA: Hemoglobin (Hb): ≤115 grams per liter (g/L) (Male[M]); ≤95 g/L (Female[F]), ≥185 g/L (M); ≥165 g/L (F), Decrease from baseline ≥20 g/L; Hematocrit: ≤0.37 volume per volume (v/v) (M); ≤0.32 v/v (F), ≥0.55 v/v (M); ≥0.5 v/v (F); Erythrocyte Count: ≥6 Tera/L; Platelet count: <100 Giga/L, ≥700 Giga/L; Leukocytes: <3 Giga/L (Non-Black [NB]); <2 Giga/L (Black [B]), ≥16 Giga/L; Neutrophils: <1.5 Giga/L (NB); <1 Giga/L (B); Lymphocytes: >4 Giga/L; Monocytes: >0.7 Giga/L; Basophils: >0.1 Giga/L; Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN ≥0.5 Giga/L).
Time Frame: From the first dose of study treatment (Day 1) up to the last dose of the study treatment + 98 days, up to 506 days
Population: The Safety population included all participants who actually received at least 1 dose or partial of a dose of the study treatment, analyzed according to the treatment participants actually received. Only those participants with data collected for specified categories are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 459 | 464
Percentage of participants
  Hb: ≤115 g/ L (M); ≤95 g/ L (F) | 6.1 | 5.0
  Hb: ≥185 g/L (M); ≥165 g/L (F) | 3.7 | 4.7
  Hb: Decrease from baseline ≥20 g/L | 9.8 | 11.4
  Hematocrit: ≤0.37 v/v (M); ≤0.32 v/v (F) | 6.1 | 5.0
  Hematocrit: ≥0.55 v/v (M); ≥0.5 v/v (F) | 23.1 | 26.5
  Erythrocyte Count: ≥6 Tera/L | 4.4 | 6.0
  Platelet count: <100 Giga/L | 0.2 | 0.6
  Platelet count: ≥700 Giga/L | 0.7 | 0.4
  Leukocytes: <3 Giga/L (NB); <2 Giga/L (B) | 0.7 | 0.6
  Leukocytes: ≥16 Giga/L | 5.2 | 4.1
  Neutrophils: <1.5 Giga/L (NB); <1 Giga/L (B): number analyzed (Participants) | 447 | 456
  Neutrophils: <1.5 Giga/L (NB); <1 Giga/L (B) | 2.7 | 1.5
  Lymphocytes: >4 Giga/L | 5.9 | 8.2
  Monocytes: >0.7 Giga/L | 65.8 | 64.9
  Basophils: >0.1 Giga/L | 28.1 | 29.5
  Eosinophils: >0.5 Giga/L or >ULN: number analyzed (Participants) | 458 | 464
  Eosinophils: >0.5 Giga/L or >ULN | 15.3 | 21.1

13. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Clinical Chemistry
Description: Blood samples were collected to determine PCSA in chemistry. PCSA criteria: Sodium: ≤129 millimoles (mmol)/L, ≥160 mmol/L; Potassium: <3 mmol/L, ≥5.5 mmol/L; Chloride: <80 mmol/L, >115 mmol/L; Glucose: ≤3.9 mmol/L and <lower limit of normal (LLN), ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted);Total cholesterol: ≥7.74 mmol/L; Creatinine kinase: >3 ULN, >10 ULN; Creatinine: ≥150 micromoles (µmol)/L (adults), ≥30% change from baseline, ≥100% change from baseline, Creatinine Clearance (CG): ≥60 - <90 milliliter per minute (mL/min), ≥30 - <60 mL/min, ≥15 - <30 mL/min, <15 mL/min; Urea nitrogen: ≥17 mmol/L; Uric acid: <120 μmol/L, >408 μmol/L; Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST): >3 ULN, >5 ULN, >10 ULN; Alkaline phosphatase (ALP): >1.5 ULN; Total bilirubin (TB): >1.5 ULN, >2 ULN; ALT and TB: ALT >3 ULN and Bilirubin > 2 ULN; Direct bilirubin (DB) and TB: DB >35% Bilirubin and Bilirubin >1.5 ULN; Albumin: ≤25 g/L.
Time Frame: From the first dose of study treatment (Day 1) up to the last dose of the study treatment + 98 days, up to 506 days
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 459 | 464
Percentage of participants
  Sodium: ≤129 mmol/L | 1.7 | 1.9
  Sodium: ≥160 mmol/L | 0 | 0.2
  Potassium: <3 mmol/L | 0.4 | 0.4
  Potassium: ≥5.5 mmol/L | 11.3 | 10.8
  Chloride: <80 mmol/L | 0 | 0.2
  Chloride: >115 mmol/L | 0 | 0.2
  Glucose: ≤3.9 mmol/L and <LLN | 7.0 | 6.5
  Glucose: ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | 7.6 | 8.8
  Total cholesterol: ≥7.74 mmol/L | 6.1 | 4.3
  Creatinine kinase: >3 ULN | 2.2 | 3.9
  Creatinine kinase: >10 ULN | 0 | 0
  Creatinine: ≥150 µmol/L | 2.6 | 3.0
  Creatinine: ≥30% change from baseline | 20.3 | 19.2
  Creatinine: ≥100% change from baseline | 0.7 | 2.4
  CG: ≥60 - <90 mL/min | 36.4 | 39.0
  CG: ≥30 - <60 mL/min | 18.5 | 16.8
  CG: ≥15 - <30 mL/min | 0 | 0.9
  CG: <15 mL/min | 0.2 | 0.4
  Urea nitrogen: ≥17 mmol/L | 0.2 | 0.4
  Uric acid: <120 μmol/L | 0 | 0.4
  Uric acid: >408 μmol/L | 37.7 | 39.7
  ALT: >3 ULN | 1.5 | 0.4
  ALT: >5 ULN | 0.2 | 0
  ALT: >10 ULN | 0 | 0
  AST: >3 ULN | 0.2 | 0.4
  AST: >5 ULN | 0 | 0.2
  AST: >10 ULN | 0 | 0
  ALP: >1.5 ULN | 3.9 | 2.8
  TB: >1.5 ULN | 0.9 | 2.2
  TB: >2 ULN | 0.2 | 0
  ALT and TB: ALT >3 ULN and Bilirubin > 2 ULN | 0.2 | 0
  DB and TB: DB >35% Bilirubin and Bilirubin >1.5 ULN: number analyzed (Participants) | 22 | 36
  DB and TB: DB >35% Bilirubin and Bilirubin >1.5 ULN | 4.5 | 5.6
  Albumin: ≤25 g/L | 0.2 | 0.4

14. Secondary Outcome: Percentage of Participants With Abnormal Results for Urine Protein in Urinalysis
Description: Urine dipstick samples were collected to determine the significant abnormalities in urine protein.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 24, 36, 52 and 64
Population: The Safety population included all participants who actually received at least 1 dose or partial of a dose of the study treatment, analyzed according to the treatment participants actually received. Only those participants with data collected at specified timepoints are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 462 | 469
Percentage of participants
  Baseline (Day 1) | 5.0 | 6.2
  Week 4: number analyzed (Participants) | 452 | 456
  Week 4 | 4.1 | 4.9
  Week 8: number analyzed (Participants) | 443 | 452
  Week 8 | 3.7 | 5.3
  Week 12: number analyzed (Participants) | 440 | 450
  Week 12 | 4.5 | 6.4
  Week 24: number analyzed (Participants) | 444 | 447
  Week 24 | 3.9 | 4.5
  Week 36: number analyzed (Participants) | 434 | 436
  Week 36 | 3.9 | 4.5
  Week 52: number analyzed (Participants) | 421 | 422
  Week 52 | 5.0 | 6.6
  Week 64: number analyzed (Participants) | 384 | 403
  Week 64 | 4.5 | 5.5

15. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) to Dupilumab
Description: Plasma samples were collected to evaluate antibodies to dupilumab. Pre-existing immunoreactivity is defined as an ADA positive response in the assay at baseline with all post-treatment ADA results negative, or an ADA positive response at baseline with all post-treatment ADA responses less than 4-fold over baseline titer levels. Treatment-emergent response is defined as a positive response in the ADA assay post first dose, when baseline results are negative or missing. Treatment-boosted response is defined as an ADA positive response in the assay post first dose that is greater-than or equal to 4-fold over baseline titer levels, when baseline results are positive.
Time Frame: Up to Week 52
Population: The ADA population included all participants in the safety population who had at least 1 reportable ADA result after first dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 452 | 461
Participants
  Pre-existing immunoreactivity | 6 | 4
  Treatment-emergent ADA response | 11 | 47
  Treatment-boosted ADA response | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs, SAEs, all-cause mortality (deaths) were collected from the first dose of study treatment (Day 1) up to the last dose of the study treatment + 98 days, up to 506 days.
Description: Analysis was performed on the Safety population. 1 participant was exposed to different treatment other than planned (was allocated to placebo arm but inadvertently received dupilumab 300 mg q2w on Day 113). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.
Arm/Group | Placebo | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 8/464 | 14/469
Serious Adverse Events (participants affected / at risk) | 79/464 | 65/469
Other Adverse Events (participants affected / at risk) | 120/464 | 125/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=464) | Dupilumab 300 mg q2w (N=469)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Colitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 5 (5) | 3 (3)
Covid-19 Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 1 (1) | 1 (1)
Nasal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 9 (10)
Pneumonia Bacterial (Infections and infestations) | 2 (2) | 2 (3)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Pseudomonal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Vocal Cord Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Postinfarction Angina (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (2) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 40 (47) | 25 (35)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Sudden Cardiac Death (General disorders) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 2 (2) | 2 (2)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=464) | Dupilumab 300 mg q2w (N=469)
Covid-19 (Infections and infestations) | 36 (38) | 45 (45)
Nasopharyngitis (Infections and infestations) | 28 (31) | 32 (39)
Headache (Nervous system disorders) | 29 (46) | 37 (72)
Accidental Overdose (Injury, poisoning and procedural complications) | 33 (35) | 31 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-10-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT04456673/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT04456673/SAP_001.pdf